CLINICAL TRIAL: NCT01057576
Title: The Effect of Artemisia Dracunculus L. on Insulin Sensitivity in Obese, Insulin-Resistant Human Subjects
Brief Title: Safety and Efficacy Study of Tarragon on Insulin Action in Humans
Acronym: 5011
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, William Cefalu, MD, Principal Investgator, Pennington Biomedical Research Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PBRC 26006
Record Dates: First submitted 2010-01-25; First posted 2010-01-27 (Estimated); Last update posted 2016-04-08 (Estimated); Status verified 2016-04

CONDITIONS: Obesity
Keywords: bioactives; insulin; botanicals
MeSH Terms: conditions — Obesity; Insulin Resistance

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PMI 5011 (Experimental): An experimental group randomized to PMI 5011
  Interventions: Dietary Supplement: An alcoholic extract of Artemisia dracunculus L.
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: An alcoholic extract of Artemisia dracunculus L. — capsule, daily dosing
  Arms: PMI 5011
Other: Placebo — capsule, daily dosage
  Arms: Placebo

SUMMARY:
Specific compounds in plants have been proposed to enhance human metabolism. The hypothesis of the study was to evaluated the effect of an extract of Russian tarragon and to determine is compounds in the plant can be measured in the serum of human subjects and whether the compound may improve human metabolism as suggested in animal studies.

DETAILED DESCRIPTION:
Artemisia dracunculus L., often called Russian tarragon, is a wild specie and a close relative of common cooking tarragon (known as French tarragon or Artemisia dracunculus sativa or dracunculoides). Artemisia and, more specifically, Artemisia dracunculus, have a storied history of medicinal use in humans, particularly for treatment of diabetes. The Artemisia dracunculus extract described in this project as PMI-5011 was originally identified from a screening of extracts for hypoglycemic activity in diabetic mice as the most promising candidate for the development of a nutritional supplement for diabetes. The active compounds in the preparation are believed to be members of the sesquiterpene, lactone or flavanoid groups, of which the Artemisia family is well known. Preliminary data from our laboratory suggests that PMI-5011 may have significant effects to improve carbohydrate metabolism by enhancing molecular events of insulin action in skeletal muscle.

PMI-5011 is an herbal botanical dietary supplement prepared from Artemisia dracunculus L. (Russian Tarragon) to help maintain normal blood glucose concentrations. PMI-5011 is an ethanolic extract from fresh herb grown in standardized hydroponic conditions for maximum consistency and nutritional content. Artemisia is a large family of herbs with a rich history of safe medicinal and culinary use. PMI-5011 is able to significantly decrease blood glucose concentrations in Streptozotocin-induced diabetic mice and in genetically diabetic KK-Ay mice. The preparation does not, however, decrease blood glucose concentrations in non-diabetic mice or rats. The historical use of the plant and its extract suggest that it is safe and its non-toxicity has been confirmed with acute and chronic toxicity studies and non-mutagenicity confirmed with AMES testing. PMI-5011 may have several modes of action leading to its ability to decrease blood glucose concentrations in diabetic animals, suggesting it is comprised of several different nutrients that act synergistically. Some in vitro activities of PMI-5011 include the modulation of GLP-1 binding to its receptor and the stimulation of insulin-mediated glucose uptake into cultured skeletal muscle cells. PMI-5011 also decreases the expression of PEPCK in the liver of diabetic animals and may decrease hepatic glucose output as a result. Recently, in an in vitro assay identified that PMI 5011 may have potent effects to reduce phosphastase activities and thereby promote insulin sensitivity.

The overall objective of the study was to evaluate the effect of a high does of PMI 5011 in obese insulin resistant, yet non-diabetic subjects. The study is a double-blind, randomized, placebo-controlled, pilot study in which subjects will be randomized to receive either placebo or PMI-5011 (4 500mg caps/TID) for a total of 3 weeks of treatment. Each subject will continue on the same dosage of PMI-5011 or matching placebo for the entire duration of treatment.

For this pilot trial, a precise technique (hyperinsulinemic-euglycemic clamps) will be used to assess insulin sensitivity.

ELIGIBILITY:
• Criteria for Inclusion

Men and women with obesity and meeting all criteria listed below will be included in the study:

* Subjects >30 years of age
* Subjects not currently treated with diabetes medication
* Fasting blood glucose at time of screening of less than 126mg/dl
* Subjects with a Body Mass Index (BMI) > 32 and <45.
* Written Informed Consent obtained PRIOR to performing any screening tests or study procedures.

  • Exclusion Criteria
* Subjects with a prior history of Type 2 diabetes.
* Women who are pregnant or who are lactating.
* Women of childbearing potential who are not using an effective method of birth control
* Type 1 diabetes.
* Subjects who are currently on thiazolidinediones (rosiglitazone or pioglitazone) or who have taken these agents in the previous 12 weeks.
* Subjects who are on concomitant therapy with glucocorticoids (except topical or inhalant glucocorticoids).
* Subjects with a history or evidence of significant gastrointestinal dysfunction
* Subjects who are taking concomitant therapy with medications known to be nephrotoxic, such as aminoglycosides, methicillin, and cyclosporin.
* Subjects who have evidence of clinically significant renal dysfunction or disease
* Subjects with clinically significant cardiovascular dysfunction and/or history
* Subjects who have evidence within the preceding 6 months of hepatic disease or dysfunction; hepatitis; jaundice; cirrhosis.
* Subjects with clinically significant pulmonary, neurologic, hematologic, immunologic, neoplastic or metabolic disease.
* Subjects with evidence or recurrence of malignancy within the past five years, other than excised basal cell carcinoma.
* Subjects for whom surgery is anticipated during the study period.
* Subjects with an history of substance abuse or alcoholism within the past 5 years, or significant psychiatric disorder that would interfere with the subject's ability to complete the study.
* Subjects who have donated blood during the month prior to study entry or planned during the study.
* Subjects who have participated in other studies using an investigational drug during the preceding 3 months.
* Subjects who are current smokers or have smoked within the previous 6 months. No smoking will be allowed during the study.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2006-03; Primary Completion 2007-03 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Insulin sensitivity | at study completion

SECONDARY OUTCOMES:
plasma abundane of bioactives | at study completion

CONTACTS AND LOCATIONS:
Overall Officials: William T Cefalu, MD, Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States